CLINICAL TRIAL: NCT01361646
Title: Safety, Tolerability and Pharmacokinetic/Pharmacodynamic Characteristics of LC350189
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-GDCL001
Record Dates: First submitted 2011-05-19; First posted 2011-05-27 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Hyperuricemia; Gout
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- LC350189 (Experimental)
  Interventions: Drug: LC350189
- Febuxostat (Active Comparator)
  Interventions: Drug: LC350189
- Placebo (Placebo Comparator)
  Interventions: Drug: LC350189

INTERVENTIONS:
Drug: LC350189 — Single Ascending Dose: 10, 25, 50, 100, 200, 400, 600mg Multifle Ascending Dose: 100, 200, 400, 600, 800mg

SUMMARY:
This will be a dose block-randomized, double-blind, active and placebo controlled, single and multiple dosing, dose-escalation study to evaluate tolerability, safety and pharmacokinetic / pharmacodynamic characteristics. Adverse events, physical examinations, vital signs, ECG and laboratory tests will be conducted for safety/tolerability evaluation and serial blood samples and urine collections for pharmacokinetic and pharmacodynamic evaluations will be conducted at specified time points.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 20 and 50 years at screening
2. Subjects with Body Mass Index (BMI) between 18.0 (inclusive) and 27.0 kg/m2 (exclusive); and a total body weight between 55 kg (inclusive) and 90 kg (exclusive). ☞ BMI (kg/m2) = body weight (kg)/ {height (m)}2.
3. Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB) - approved informed consent prior to performing any of the screening procedures.
4. Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the laboratory reference ranges for the relevant laboratory tests

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Adverse events of LC350189 | 7 days(plus or minus 1 day)

SECONDARY OUTCOMES:
Cmax | 3 days
AUC | 3days
Tmax | 3days

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea